CLINICAL TRIAL: NCT00987142
Title: A Comparative Open-Label Multicentre Clinical Trial To Assess The Efficacy And Safety Of A New Therapy With Cultured Chimeric Skin For The Treatment Of Skin Lesions In Patients With Epidermolysis Bullosa
Brief Title: Trial To Assess Efficacy Of A Chimeric Skin In Patients With Epidermolysys Bullosa
Acronym: TCEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX501/TCEB
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: EPIDERMOLYSIS BULLOSA
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CX501 (Experimental): Cultured chimeric skin
  Interventions: Drug: CX501
- Non adherent dressing (Active Comparator): Occlusive non adherent dressing
  Interventions: Device: Occlusive non adherent dressing

INTERVENTIONS:
Drug: CX501 — Cultured chimeric skin
  Arms: CX501
Device: Occlusive non adherent dressing — Application of an occlusive non adherent dressing in the skin donor site
  Arms: Non adherent dressing

SUMMARY:
A phase II, comparative, open label, prospective, multicentre clinical trial where each patient will undergo two procedures; implant of a patch of cultured chimeric skin (experimental therapy) in a half of the skin lesion and an occlusive non-adherent dressing (control) in the other half for 12 months of follow-up in two Spanish centres.

DETAILED DESCRIPTION:
Reconstruction of interdigital commisures in patients with severe skin syndactyly using laminar grafts that will be uniformly and systematically taken with an electrical or compressed air dermatome on an aseptic area and with the same extent and depth in microns in all patients.

Immediately after the surgical procedure, a patch of cultured chimeric skin (experimental therapy) will be implanted in a half of the skin defect of the patient, and an occlusive non - adherent dressing (control) will be implanted in the other half.

Patients will initially be followed up every two days until epithelisation occurs (approximately 21 days after surgery) and at 3,8,and 12 months of follow-up.

ELIGIBILITY:
Inclusion criteria:

* Patients of both sexes over 28 days of age.
* Patients with recessive dystrophic epidermolysis bullosa diagnosed by clinical and historical criteria with severe skin syndactyly in whom reconstructive surgery is indicated.
* Patients whose legal guardians have given written informed consent for participation in the study before any study procedure is performed.
* Patients aged ≥ 12 years who have given written informed consent for participation in the study before any study procedure is performed.

Exclusion criteria:

* Women of childbearing age not using effective contraceptive methods (oral contraception)
* Pregnant or nursing women
* Documented or suspected hypersensitivity to any of the therapeutic agents included in the study, including anaesthetic drugs.
* Patients with a history of malignant tumor in the past 5 years
* Patients with a diagnosis of active tuberculosis at the time of recruitment
* Patients with prior positive markers for any of the following pathogens: hepatitis b and c, hiv-1 and hiv-2
* Patients with a history of clinically relevant hepatic, gastrointestinal, haematological, pulmonary, or neurological disease no directly related to epidermolysis bullosa.
* Any other medical condition which, in the investigator´s judgment, might interfere with optimal participation in the study or involve a significant risk for the patient.
* Alcoholism, drug addiction, psychiatric disorders, or other factors present in legal guardians which,in the investigator´s judgment may complicate patient participation in the study.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Time to epithelization | 21 days

SECONDARY OUTCOMES:
Fibroblast persistence | 3, 8 and 12 months
Incidence of Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos López, MD, Principal Investigator — Hospital La Paz
Locations (2):
- Spain (2):
  - Fundación Mir-Mir, Barcelona
  - Hospital La Paz, Madrid